CLINICAL TRIAL: NCT03704493
Title: The Impact of Virtual Group Motivation on the Performance and Comfort of Patients in Exercise Treadmill Testing: A Randomized, Open Label Trial
Brief Title: Virtual Group Motivation in Exercise Treadmill Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Urs Hufschmid, Head of Cardiology, Principal Investigator, Kantonsspital Baden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ErgoTrial
Record Dates: First submitted 2018-09-10; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Exercise Test
Keywords: Exercise testing; coronary artery disease; virtual group motivation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The intervention consists of a video shown to the patient while exercising on the treadmill. It shows 5 amateur runners running across woods and fields. The group is film form behind giving the patient the impression of running within the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Image Group (No Intervention): The patients were looking at a static image of a lavender flower while exercising on the treadmill.
- Video Group (Experimental): The patients were watching a video of a group of amateur runners while exercising on the treadmill.
  Interventions: Diagnostic Test: Video Group

INTERVENTIONS:
Diagnostic Test: Video Group — A video of a group of five amateur runners running along woods and fields. The group was filmed from behind to give the patient the impression of running within the group.
  Arms: Video Group

SUMMARY:
Exercise stress testing is the most frequently used clinical tool for assessment of coronary artery disease. To ensure a high validity of the results, a good Patient compliance is crucial. The aim of this study is to examine the effects of a virtually presented exercise group on the perceived comfort and the exercise capacity of patients during classical treadmill exercise testing. The investigators hypothesis is, that a virtually presented running group will increase the comfort of patients and their exercise capacity.

DETAILED DESCRIPTION:
108 Patients were randomized in an open label trial 1:1 to either exercise treadmill testing while watching a static image of a flower (image group) or to exercise treadmill testing while watching a video of 5 amateur runners, running across and fields, giving the patient the impression of running within the group (video group). After the exercise test patients were asked to score their perceived comfort level and achieved level of their subjective physical limit on a 10 point scale.

Standard exercise treadmill parameters, as well as baseline demographic data were recorded of each patient. Patients with missing data was excluded of the analysis.

Statistic analysis was performed with t-test for normally distributed data and Wilcoxon-Mann-Whitney-Test for non-normal data.

ELIGIBILITY:
Inclusion Criteria:

* indication for exercise stress testing

Exclusion Criteria:

* any contraindication for exercise stress testing
* unability of performing an exercise treadmill test
* recent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2014-09-26 (Actual); Study Completion 2014-09-26 (Actual)

PRIMARY OUTCOMES:
Patients' performance | Day of Exercise Testing
  Patients' performance in metabolic equivalents percentage of age predicted maximum
Patients' comfort | Day of Exercise Testing
  Subjective level of comfort of patient during the exercise test rated on a 10 point scale. Scale ranges from 1 to 10. 10 indicates that the patient felt absolutely comfortable during the test, 1 indicates that the patient did not feel comfortable at all.

SECONDARY OUTCOMES:
Exercise test duration | Day of Exercise Testing
  Exercise test duration in min:sec
Age predicted heart rate | Day of Exercise Testing
  achieved percentage of age predicted heart rate
physical limits | Day of Exercise Testing
  Achieved subjective level of physical limit rated on a 10 point scale. Scale ranges from 1 to 10, 10 indicates that the patient subjectively reached his physical Limit, 1 indicates that the patient did not reach his physical limit at all. The higher the value the more did the patient reach his physical limit (the better the outcome).
rate pressure product increase | Day of Exercise Testing
  increase of the rate pressure product during the test

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Hans Beer, Prof., Study Director — Head of the Department of Internal Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilzeck VC, Hufschmid J, Bischof L, Hansi C, Nagele MP, Beer JH, Hufschmid U. A significant increase in exercise test performance with virtual group motivation: a randomised open-label controlled trial. Swiss Med Wkly. 2020 Jul 15;150:w20287. doi: 10.4414/smw.2020.20287. eCollection 2020 Jul 13. PMID 32725609